CLINICAL TRIAL: NCT02217566
Title: Abiraterone Acetate in Patients With Metastatic Castration-Resistant Prostate Cancer, Chemo-Naive, Who Received a Prior Diethylstilbestrol Therapy
Brief Title: Study of Abiraterone Acetate in Participants With Metastatic Castration-Resistant Prostate Cancer (mCRPC), Chemo-Naive, Who Received a Prior Diethylstilbestrol Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR103352; 212082PCR2036 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic neoplasms; Diethylstilbestrol therapy; Abiraterone acetate; Prednisone; Androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Abiraterone Acetate (Experimental): Participants will receive abiraterone acetate 1000 milligram (mg) orally once daily along with prednisone 5 mg orally once daily and androgen deprivation therapy (ADT) as per Investigator's discretion until prostate-specific Antigen (PSA) progression, clinical progression, consent withdrawal, or the occurrence of unacceptable toxicity.
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone; Drug: Androgen deprivation therapy (ADT)

INTERVENTIONS:
Drug: Abiraterone acetate — Participants will receive abiraterone acetate 1000 mg (4*250 mg tablets) orally once daily until PSA progression, clinical progression, consent withdrawal, or the occurrence of unacceptable toxicity.
  Other Names: ZYTIGA®; JNJ-212082
Drug: Prednisone — Participants will prednisone 5 mg orally once daily from Day 1 of Cycle 1 and continues until PSA progression, clinical progression, consent withdrawal, or the occurrence of unacceptable toxicity.
Drug: Androgen deprivation therapy (ADT) — Participants will remain on a stable regimen of ADT, that is, luteinizing hormone-releasing hormone (LHRH) agonists including leuprolide acetate and goserelin acetate as per Investigator's discretion.

SUMMARY:
The purpose of this study is to evaluate the efficacy, based on prostate-specific antigen (PSA) progression, of abiraterone acetate in participants with metastatic (spread of cancer cells from one part of the body to another) castration (any action, surgical, chemical, or otherwise, by which a male loses the functions of the testes) resistant prostate cancer (cancer in prostrate; a gland that makes fluid that aids movement of sperm) (mCRPC), chemo-naive (treatment of cancer is not done using drugs), who received a prior diethylstilbestrol therapy (DES).

DETAILED DESCRIPTION:
This is a Phase 2, multinational (when medical research study takes place in more than one country), multicenter (when more than one hospital or medical school team work on a medical research study), open-label (all people know the identity of the intervention), and single arm study to determine benefits of abiraterone acetate and low-dose prednisone to androgen deprivation therapy (ADT) in mCRPC participants who failed to prior DES therapy. The study will consist of a Screening Phase of up to 28 days before enrollment; a PSA Evaluation Phase; and a Follow-up Phase of up to 24 months. Each cycle of abiraterone therapy will be of 28 days. Participants will receive 1000 milligram (mg) abiraterone acetate orally once daily plus prednisone 5 mg orally once daily plus stable regimen of ADT (luteinizing hormone-releasing hormone [LHRH] agonists) as per Investigator's discretion. Treatment will continue until PSA progression, clinical progression, consent withdrawal, or the occurrence of unacceptable toxicity. Efficacy will primarily be assessed by time to PSA progression. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology
* Prior therapy with diethylstilbestrol (DES) for castration resistant prostate cancer. Participants should demonstrate evidence of progression on DES or evidence of grades 3/4 toxicities on DES
* Metastatic disease documented by positive bone scan or metastatic lesions on computerized tomography (CT) or magnetic resonance imaging (MRI)
* May have received prior androgen blockage (bicalutamide or flutamide) but must have been discontinued for least 28 days
* Ongoing androgen deprivation therapy (ADT) (luteinizing hormone-releasing hormone [LHRH] agonist or orchiectomy), with serum testosterone level of less than 50 nanogram per deciliter (1.7 nanomole per liter) and eligible participants must maintain ADT

Exclusion Criteria:

* Active infection or other medical condition that would make prednisone use contraindicated
* Any chronic medical condition requiring a higher systemic dose of corticosteroid than 5 milligram (mg) prednisone per day
* Pathological finding consistent with small cell carcinoma of the prostate
* Known brain metastasis
* Has had prior cytotoxic chemotherapy or biologic therapy for the treatment of metastatic castration-resistant prostate cancer (mCRPC)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- Brazil (4):
  - Porto Alegre
  - Rio de Janeiro
  - Santo André
  - São Paulo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 46 participants were enrolled into the study and were treated with abiraterone acetate and prednisone. Out of 46 participants, 6 did not fulfill all eligibility criteria and included in the safety population. Thirty-five (35) participants completed the study.
Groups:
- Abiraterone Acetate: Participants received abiraterone acetate 1000 milligram (mg) orally once daily along with prednisone 5 mg orally once daily and androgen deprivation therapy (ADT) as per Investigator's discretion until prostate-specific Antigen (PSA) progression, clinical progression, consent withdrawal, or the occurrence of unacceptable toxicity.
Period: Overall Study
Arm/Group | Abiraterone Acetate
Started | 46
Completed | 35
Not Completed | 11
Not completed — Lost to Follow-up | 2
Not completed — Death | 3
Not completed — Early study termination | 6

BASELINE CHARACTERISTICS:
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (7.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Pacific Islander | 1
  Black or African/South American | 7
  Other | 1
  White/Caucasian | 37
Region of Enrollment [Count of Participants; unit: Participants]
  BRAZIL | 46

OUTCOME MEASURES:

1. Primary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: Time to PSA progression was calculated from date of enrollment to the date of first documentation of PSA progression. As per Prostate Cancer Clinical Trials Working Group (PCWG2) criteria, PSA progression was defined as greater than or equal to (>=) 25 percent (%) and >=2 nanogram/milliliter (ng/mL) after 12 weeks (in case of no decline in PSA from Baseline), or first PSA increase that is >=25% and >=2 ng/mL above the nadir, and which was confirmed by a second value 3 or more weeks later (in case of decline of PSA from Baseline).
Time Frame: Up to 2 years
Population: The efficacy population included all eligible participants who received at least one dose of any study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 40
Months | 7.3 [5.6 to 10.0]

2. Secondary Outcome: Percentage of Participants Who Achieved Prostate-Specific Antigen (PSA) Response
Description: The PSA response according to Prostate Specific Antigen Working Group 3 criteria was defined as at least 50% decrease in PSA level from Baseline.
Time Frame: Week 12 to any time up to 2 years
Population: The efficacy population included all eligible participants who received at least one dose of any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 40
Percentage of participants | 57.50 [27.0 to 59.1]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from date of the first dose of abiraterone acetate to the date of death due to any cause. For participants who did not die until the time of analysis, survival time was censored at the time of last contact alive.
Time Frame: Up to 4 years
Population: The efficacy population included all eligible participants who received at least one dose of any study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 40
Months | 29.6 [16.10 to NA] — Here, NA signifies that the number of participants with events was not sufficient to provide upper confidence limit estimate for median as curve representing upper confidence limits for survival function lies above 0.50.

4. Secondary Outcome: Percentage of Participants With Pain Progression as Assessed by Brief Pain Inventory - Short Form (BPI-SF) - Pain Severity Score
Description: The BPI-SF is a publicly available instrument to assess the pain and includes severity and interference scores. BPI-SF is an 11-item self-report questionnaire that is designed to assess the severity and impact of pain on daily functions of a participant. Pain severity score is a mean value for BPI-SF questions 3, 4, 5 and 6 (questions inquiring about the extent of pain, where the extent is ranked from 0 [no pain] to 10 [pain as bad as you can imagine]). Pain severity progression was defined as an increase in score of 30% or greater from baseline without decrease in analgesic use.
Time Frame: Up to 2 years
Population: The efficacy population included all eligible participants who received at least one dose of any study drug and with at least 2 BPI-SF assessments after baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 36
Percentage of participants | 19.44

5. Secondary Outcome: Percentage of Participants With Pain Progression as Assessed by Brief Pain Inventory - Short Form (BPI-SF) - Pain Interference Score
Description: The BPI-SF is a publicly available instrument to assess the pain and includes severity and interference scores. BPI-SF is an 11-item self-report questionnaire that is designed to assess the severity and impact of pain on daily functions of a participant. Pain interference score is mean value for the 7 BPI-SF questions (questions inquiring about the extent of interference with activities by pain) where the extent is ranked from 0 (does not interfere) to 10 (completely interferes). Pain interference progression was defined as an increase in score of 50% or greater from baseline without decrease in analgesic use.
Time Frame: Up to 2 years
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 33
Percentage of participants | 15.15

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant who will receive study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly.
Time Frame: Up to 4 years
Population: The safety population included all participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 46
Participants
  Participants with AEs | 45
  Participants with SAEs | 11

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: Safety population included all participants who received at least 1 dose of any study drug.
Arm/Group | Abiraterone Acetate
All-Cause Mortality (participants affected / at risk) | 3/46
Serious Adverse Events (participants affected / at risk) | 11/46
Other Adverse Events (participants affected / at risk) | 45/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=46)
Anaemia (Blood and lymphatic system disorders) | 1
Cardiac Failure (Cardiac disorders) | 2
Cardio-Respiratory Arrest (Cardiac disorders) | 1
Amaurosis (Eye disorders) | 1
Gastrointestinal Obstruction (Gastrointestinal disorders) | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Cystitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1
Ulna Fracture (Injury, poisoning and procedural complications) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Spinal Cord Compression (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=46)
Anaemia (Blood and lymphatic system disorders) | 13
Eosinophilia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Atrial Fibrillation (Cardiac disorders) | 1
Atrioventricular Block (Cardiac disorders) | 1
Bundle Branch Block Left (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Conjunctival Haemorrhage (Eye disorders) | 1
Eye Pain (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Ocular Hyperaemia (Eye disorders) | 1
Papilloedema (Eye disorders) | 1
Vision Blurred (Eye disorders) | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 3
Abdominal Pain Lower (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 8
Abdominal Wall Haematoma (Gastrointestinal disorders) | 1
Anal Incontinence (Gastrointestinal disorders) | 1
Anorectal Discomfort (Gastrointestinal disorders) | 1
Aphthous Ulcer (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 9
Diverticulum (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 11
Odynophagia (Gastrointestinal disorders) | 2
Proctalgia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 8
Chest Pain (General disorders) | 4
Face Oedema (General disorders) | 1
Fatigue (General disorders) | 15
Influenza Like Illness (General disorders) | 4
Localised Oedema (General disorders) | 1
Malaise (General disorders) | 3
Mucosal Inflammation (General disorders) | 1
Oedema Peripheral (General disorders) | 9
Pyrexia (General disorders) | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Anal Abscess (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 7
Nasopharyngitis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Strongyloidiasis (Infections and infestations) | 1
Subcutaneous Abscess (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 7
Eye Injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 4
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1
Joint Injury (Injury, poisoning and procedural complications) | 1
Sciatic Nerve Injury (Injury, poisoning and procedural complications) | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 2
Blood Alkaline Phosphatase Increased (Investigations) | 3
Blood Bilirubin Increased (Investigations) | 2
Blood Creatinine Increased (Investigations) | 2
Blood Lactate Dehydrogenase Increased (Investigations) | 1
Blood Pressure Increased (Investigations) | 1
ECG Electrically Inactive Area (Investigations) | 1
International Normalised Ratio (Investigations) | 1
Platelet Count Decreased (Investigations) | 2
Weight Decreased (Investigations) | 6
Weight Increased (Investigations) | 1
White Blood Cell Count Decreased (Investigations) | 3
Decreased Appetite (Metabolism and nutrition disorders) | 11
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 17
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Metabolic Acidosis (Metabolism and nutrition disorders) | 1
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 21
Bone Pain (Musculoskeletal and connective tissue disorders) | 2
Coccydynia (Musculoskeletal and connective tissue disorders) | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck Pain (Musculoskeletal and connective tissue disorders) | 5
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 12
Spinal Pain (Musculoskeletal and connective tissue disorders) | 2
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 11
Motor Dysfunction (Nervous system disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 4
Syncope (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 9
Haematuria (Renal and urinary disorders) | 6
Lower Urinary Tract Symptoms (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Urethral Haemorrhage (Renal and urinary disorders) | 1
Urethral Pain (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 2
Gynaecomastia (Reproductive system and breast disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 3
Penile Burning Sensation (Reproductive system and breast disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Tracheal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Upper Respiratory Tract Irritation (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hyperaemia (Vascular disorders) | 2
Hypertension (Vascular disorders) | 19
Hypotension (Vascular disorders) | 2
Shock (Vascular disorders) | 1
Varicose Vein (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT02217566/Prot_SAP_000.pdf